CLINICAL TRIAL: NCT01514916
Title: Evaluation of a Mechanical System (Vascular Join) Facilitating Arterial Anastomoses During Peripheral Vascular Surgery (Bypass).
Brief Title: New Anastomotic Device for End to End Vascular Anastomosis in the Treatment of Peripheral Vascular Disease
Acronym: VJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ab Medica Spa (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK VD 64/08
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Peripheral Vascular Disease; Femoral Occlusive Disease; Femoropopliteal Occlusive Disease; Aortoiliac Atherosclerosis
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: mechanical anastomosis without suture — The Vascular Join device is intended to be used to create sutureless end-to-end anastomosis between an artery and a venous or synthetic graft conduit. Any type of e-PTFE and Dacron conduits can be used.

SUMMARY:
The medical device "Vascular Join" represents a new anastomotic technology that should reduce the inter-surgeons variability in anastomosis construction and increase the performances in terms of results. It allows a perfect mechanical anastomosis without suture, avoiding the disadvantages of operation length and difficulty of the act, thrombosis, clamping and embolism. The "Vascular Join" creates automatically the connection between the vein or prosthesis at both ends and bridging the artery while preventing the passage of the needle and suture through the vessel wall and clamping pressure. This makes it very easy to construct a vascular anastomosis using the endoscopic technique less traumatic for the patient, lessen the pain of the patient, thereby reducing health care costs by reducing the length of hospital stay.

No part of the device is in contact with the patient's blood because the whole system remains in the thickness of the arterial wall and outside the vessel. Thus, the formation of intimal hyperplasia is greatly diminished and the risk of occlusion of the anastomosis is less than the currently available risk when a suture is used. This risk is shown by studies on animals in labs, with a mean follow up of 12 months. The Vascular Join creates a perfect congruence of anastomosed vessels because it allows a perfect match between each vascular tunic.

The medical device Vascular Join has been designed in order to:

* Reduce the suture time;
* Reduce the risk of occlusion of vein after the surgical process;
* Avoid the contact risk between the external material steel (surgical needle) and blood;
* Standardize the quality of anastomoses independently of the skill of the surgeon.

DETAILED DESCRIPTION:
The Vascular Join consists of two symmetrical parts, called Vessel Rings, each of which is fixed to the extremity of the two conduits being joined together. A third ring, called Coupler Ring, keeps the two rings together with a snap-on system and guarantees the continuity of the severed conduit in an end-to-end configuration. Each ring is made within a cylinder-type steel AISI 316L. The circular shape of the Vessel rings, the inner part in particular, provides a natural physiologic vascular reconstruction reducing the risk of thrombosis and myointimal hyperplasia at the anastomotic site.

We propose to evaluate the ease of use, efficiency, security of the "Vascular Join" and long-term results (6 months) in patients with peripheral vascular disease requiring vascular bypass. Each patient has a proximal anastomosis and distal anastomosis performed with the "Vascular Join". Next, measure the flow in the bypass through an ultrasonic flow meter.

The objective is to achieve a vascular bypass using the mechanical device described above and to define the incidence of major and minor vascular complications in the postoperative 7 days (or until discharge), as well as primary and secondary permeability bypass after 6 months. What we define as major vascular complications are death, stroke, acute occlusion, partial occlusion, and reoperation for redo the mechanical anastomosis. We define as minor complications residual pain, and bleeding.

In the case of partial or complete failure of the mechanical suture, the surgeon can add points of suture or performing anastomosis with the traditional technique.

After 6 months, a Doppler will allow us to compare to each patient, the morphology of the anastomoses performed with the "Vascular Join," and the permeability of the bypass. The results will be compared to historical results of primary and secondary permeability present in the literature.

The 2 main objectives of this study are to assess if the device still works after 6 months (so called device's performance) and if it is as safe as standard technique (running or interrupted suture) in terms of incidence of complications as bleeding, infection and occlusion. Simple size has therefore been calculated in terms of equivalence risk. In this case the null hypothesis specify that the success rate Pc in the standard treatment is higher than the success rate PE in the vascular join treatment by at least some amount ß.

The alternative hypothesis specifies that PC - PE < ß, which implies the 2 therapies are equivalent. The following formula provides the required number of patients for such a trial:

Ho: PC >(or =) PE + ß vs H1: PC <(or =) PE + ß . Because, taking historical data as reference, the incidence of all complications in peripheral bypasses could be as high as 50% at 6 months, the number of 30 patients was selected.

The post-operative treatment and remote monitoring of patients remained unchanged (Aspirin 100 mg/d and control angiological at 3 and 6 months).

Patient's follow-up is the same as any other patient receiving femoral artery bypass, which means physical examination and Doppler ultrasound of the bypass before the discharge, 1, 3 and 6 months after the procedure.

If the patient misses the scheduled control, the PI will apply the procedure in use at the Cardiovascular Surgery Dpt to contact him, which includes phone calls to the patient, the contact person he/her identified at the admission and to the GP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral vascular disease requiring vascular bypass (Fontaine stage 2B-3)

Exclusion Criteria:

* Pregnant women
* Patient requiring further surgery at the same time
* A patient with acute vascular occlusion.
* Hemodynamically unstable patient before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications using Vascular Join | six month
  The objective is to achieve a vascular bypass using the mechanical device Vascular Join and define the incidence of vascular complications (bleeding, infection and occlusion) in the postoperative 7 days (or until discharge), as well as primary and secondary permeability bypass after 6 months. The incidence is compared with the Vascular standard technique (running or interrupted suture).

CONTACTS AND LOCATIONS:
Overall Officials: Cosimo Puttilli, Eng., Study Director — Ab Medica Spa
Locations (1):
- Service de Chirurgie cardio-vasculaire CHUV, Lausanne, Switzerland

REFERENCES:
- [Background] Tozzi P, Borghi E, Haesler E, Siniscalchi G, Motti A, Hayoz D, von Segesser LK. Progress in cardiovascular anastomoses: will the vascular join replace Carrel's technique? Eur J Cardiothorac Surg. 2006 Sep;30(3):425-30. doi: 10.1016/j.ejcts.2006.05.029. Epub 2006 Jul 20. PMID 16859919
- [Background] Ferrari E, Tozzi P, von Segesser LK. The Vascular Join: a new sutureless anastomotic device to perform end-to-end anastomosis. Preliminary results in an animal model. Interact Cardiovasc Thorac Surg. 2007 Feb;6(1):5-8. doi: 10.1510/icvts.2006.137943. Epub 2006 Nov 20. PMID 17669755
- [Background] Tozzi P, Solem JO, Boumzebra D, Mucciolo A, Genton CY, Chaubert P, von Segesser LK. Is the GraftConnector a valid alternative to running suture in end-to-side coronary arteries anastomoses? Ann Thorac Surg. 2001 Sep;72(3):S999-1003. doi: 10.1016/s0003-4975(01)02953-8. PMID 11565736